CLINICAL TRIAL: NCT05029518
Title: A Phase 1, Randomized, Open-Label, Single-Dose, 3-Way Crossover Study to Compare the PK of Two Oral Formulations of SMP-100 and to Evaluate the Effect of Food on the Bioavailability of SMP-100 Tablets in Normal Healthy Volunteers
Brief Title: 3-Way Crossover Study to Compare the PK (Pharmokinetics) and to Evaluate the Effect of Food on the Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu SciMount Pharmatech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SciMount
Record Dates: First submitted 2021-08-22; First posted 2021-08-31 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A: SMP-100 dissolved in water administered under fasting conditions (Experimental): 12 subjects，For Treatment A, SMP-100 will be dissolved in a total of 240 mL of water and administered orally to each subjects, and a hand and mouth check will be performed to ensure consumption of the medication. Subjects will be required not to wear dentures or mouth piercing at the time of dosing. No food will be allowed from at least 10 hours before dosing until at least 4 hours post-dose.
  Interventions: Drug: SMP-100
- Treatment B: SMP-100 tablets administered under fasting conditions (Experimental): 12 subjects，For Treatment B, SMP-100 tablets will be administered to each subject with 240 mL of water and a hand and mouth check will be performed to ensure consumption of the medication. The dosing procedure must be completed within 2 minutes. In the event that subjects cannot swallow all tablets with 240 mL of water, additional water may be allowed up to a maximum total volume of 400 mL. No food will be allowed from at least 10 hours before dosing until at least 4 hours post-dose.
  Interventions: Drug: SMP-100
- Treatment C: SMP-100 tablets administered under fed conditions (Experimental): 12 subjects，For Treatment C, SMP-100 tablets will be administered to each subject with 240 mL of water and a hand and mouth check will be performed to ensure consumption of the medication. The dosing procedure must be completed within 2 minutes. In the event that subjects cannot swallow all tablets with 240 mL of water, additional water may be allowed up to a maximum total volume of 400 mL.
  After a supervised fast of at least 10 hours, subjects will be served a high-fat, high-calorie meal of approximately 800 to 1000 calories (approximately 50% of total caloric content of the meal derived from fat). This test meal should derive approximately 150, 250, and 500-600 calories from protein, carbohydrate, and fat, respectively. Subjects should start the meal approximately 30 minutes prior to drug administration. Subjects will be required to completely eat the meal in 30 minutes or less. No food will be allowed until at least 4 hours post-dose.
  Interventions: Drug: SMP-100

INTERVENTIONS:
Drug: SMP-100 — In each period, subjects will receive a single dose of SMP-100 on Day 1 (Period 1), Day 4 (Period 2), and Day 7 (Period 3), under fasting or fed conditions, followed by 48 hours of PK and safety assessments.
  Other Names: ALB-137391(a); CSTI-300; SMP-100 oral solution; SMP-100 tablet

SUMMARY:
This is a single center, Phase 1, randomized, open-label, single-dose, 3 treatment, 3-period, 6-sequence, crossover study designed to compare the PK of SMP-100 dissolved in water for oral administration with SMP-100 tablets under fasting conditions, and to evaluate the effect of food on the bioavailability of SMP-100 tablets in healthy subjects.

DETAILED DESCRIPTION:
SMP-100 is a novel serotonin receptor 3 (5-HT3) partial agonist. The compound is under development in an oral dosage form for the treatment of diarrhea-predominant irritable bowel syndrome (IBS-d). The study drug also has the potential to treat chemotherapy induced nausea and emesis and diarrhea due to carcinoid syndrome.

A single ascending dose (SAD) and multiple ascending dose (MAD) clinical study (study number SMP-100-101) evaluating the safety, tolerability, and PK profile of orally administered SMP-100 in healthy volunteers is ongoing. Regarding safety, there have been no clinically relevant abnormal vital signs, ECGs, laboratory results or SAEs.

In each period, subjects will receive a single 4 mg dose of SMP-100 on Day 1 (Period 1), Day 4 (Period 2), and Day 7 (Period 3), under fasting or fed conditions, followed by 48 hours of PK and safety assessments.

The study will include a screening visit from Day -28 to Day -2. Eligible subjects will be admitted to the clinical site on Day -1 and will be confined until completion of the assessments on Day 9. There will be a washout period of at least 72 hours between doses.

Primary objectives:

* To compare the PK of SMP-100 dissolved in water for oral administration with SMP-100 tablets under fasting conditions, following a single dose in healthy subjects.
* To evaluate the effect of a high-fat, high-calorie meal on the bioavailability of SMP-100 tablets, following a single dose in healthy subjects.

Secondary objective:

• To evaluate the safety and tolerability of two SMP-100 oral formulations when administered to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥18 and ≤59 years old at time of screening.
2. Body mass index (BMI) >18.5 and <30.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
3. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
   3. the absence of clinically significant history of constipation, diarrhea, or irregular bowel transit in the last 4 weeks.
   4. the absence of clinically significant history of irritable bowel syndrome (IBS) of any type.
   5. the absence of current or history of ischemic colitis.
   6. the absence of any other gastrointestinal disease which could interfere with the absorption of orally-administered medication.
4. Female subjects of non-childbearing potential must be:

   1. post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented follicle-stimulating hormone (FSH) levels ≥40 mIU/mL at screening; or
   2. surgically sterile (bilateral oophorectomy, hysterectomy or tubal ligation at least 3 months prior to dosing).
5. Sexually active female subjects of childbearing potential and non-sterile male subjects must be willing to use an acceptable contraceptive method throughout the study as detailed in section 11.1.
6. Willing to take off dentures or mouth piercing at the time of dosing (for Treatment A).
7. Able to understand the study procedures and provide signed informed consent form (ICF) to participate in the study.

Exclusion Criteria:

1. Any clinically significant (in the opinion of the Investigator) abnormal finding at physical examination at screening.
2. Any clinically significant (in the opinion of the Investigator) abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody at screening.
3. Positive pregnancy test or lactating female subject.
4. Positive urine drug screen, urine cotinine test, or alcohol breath test at screening or Day -1.
5. Known allergic reactions to any excipient in the formulations.
6. History of hypersensitivity to 5-hydroxytryptamine 3 receptor (5-HT3) receptor antagonists or agonists.
7. Clinically significant ECG abnormalities (Fridericia's corrected QT interval [QTcF] >450 ms for males and >470 ms for females).
8. Clinically significant vital signs abnormalities (systolic BP lower than 90 or over 160 mmHg, diastolic BP lower than 50 or over 95 mmHg, or HR less than 45 bpm) at screening.
9. Clinically significant orthostatic vital signs abnormalities such as decrease in systolic BP of 20 mmHg or higher, decrease in diastolic BP of 10 mmHg or higher, or increase in HR of 30 bpm or higher within 3 minutes after passing from a supine to a standing position.
10. History of significant drug abuse within 1 year prior to screening or use of drugs such as marijuana within 3 months prior to the screening visit or drugs such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives within 1 year prior to screening.
11. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit that exceeds 14 units of alcohol per week (1 unit = 150 mL of wine, 375 mL of mid strength beer, or 30 mL of distilled alcohol 40%).
12. Use of medications within the timeframes specified in section 11.2.
13. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing or of a biological product within 90 days prior to dosing.
14. Previous participation in a clinical research study involving the administration of SMP-100.
15. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
16. Presence of orthodontic braces or orthodontic retention wires, or any physical findings in the mouth or tongue that would be likely to interfere with successful completion of the dosing procedure.
17. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Primary PK endpoints: AUC( 0-inf) | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Area under the concentration-time curve from time zero to infinity (extrapolated)
Primary PK endpoint: AUC(0-t) | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Area under the concentration-time curve from time zero until the last observed concentration
Primary PK endpoint: Cmax | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Maximal observed concentration

SECONDARY OUTCOMES:
Secondary PK endpoint: Tmax | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Time when the maximal concentration is observed
Secondary PK endpoint: Tlag | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Time of observation prior to the first observation with a measurable (non-zero)
Secondary PK endpoint: T½ el | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Terminal elimination half-life
Secondary PK endpoint: Kel | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Elimination rate constant
Secondary PK endpoint: Cl/F | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Apparent body clearance
Secondary PK endpoint: Vz/F | pre-dose and 0.25, 0.5, 1, 1.33, 1.67, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, and 48 hours post-dose
  Apparent volume of distribution
Adverse event profile | Day -1 to Day 9
  Nature, incidence and severity of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Polasek, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, Australia